CLINICAL TRIAL: NCT01371812
Title: A Randomised, Double-blind, Placebo-controlled, Cross-over Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of GSK2239633 in Healthy Male Subjects.
Brief Title: GSK2239633 FTIH Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 114660
Record Dates: First submitted 2011-05-05; First posted 2011-06-13 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cohort 1 (Experimental): Interlocking design with Cohort 2. Single dose; treatment period over 2 days such that one subject will receive GSK2239633 and one subject will receive placebo on Day 1. The remaining subjects will be dosed on day 2 of each treatment period assuming adequate safety from Day 1. Placebo and an escalation of GSK2239633 from 150mg, to 600mg, to 1200mg and 1200mg with a FDA high fat/high calorie meal, will be administered over the 13 week long study allowing adequate washout period between doses.
  Interventions: Drug: GSK2239633; Drug: Placebo
- Cohort 2 (Experimental): Interlocking design with Cohort 1. Single dose; treatment period over 2 days such that one subject will receive GSK2239633 and one subject will receive placebo on Day 1. The remaining subjects will be dosed on day 2 of each treatment period assuming adequate safety from Day 1. Placebo and an escalation of GSK2239633 from 300mg, to 900mg, and 1500mg, will be administered over the 13 week long study allowing adequate washout period between doses.
  Interventions: Drug: GSK2239633; Drug: Placebo

INTERVENTIONS:
Drug: GSK2239633 — Drug will be orally administered at the doses and time points detailed in the 'arms' section.
Drug: Placebo — Placebo will be orally administered to 4 subjects in each treatment period of each cohort.

SUMMARY:
The purpose of this first time into human study is to investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of GSK2239633 in healthy male subjects.

DETAILED DESCRIPTION:
GSK2239633 is a human chemokine receptor 4 (CCR4) antagonist with a novel anti-inflammatory profile acting mainly on a subset of Th2 cells, with potential for the oral treatment of all severities of asthma. Inhibition of the CCR4 receptor represents a target for asthma because of the potential to inhibit Th2 cell chemotaxis and the subsequent effects of limiting Th2 cell involvement in both the acute and chronic inflammatory response. Recent data in man suggests that the CCR4 receptor ligands (thymus and activation-regulated chemokine (TARC) and macrophage-derived chemokine (MDC)) may be important in asthma and in the development of Allergic Bronchopulmonary Aspergillosis (ABPA). This will provide a unique opportunity to differentiate GSK2239633 significantly from other oral non-steroidal asthma treatments. This study is the first administration of oral GSK2239633 in humans. Two alternating cohorts of 12 subjects will receive 3 single, ascending doses of oral GSK2239633 or placebo. In addition, one cohort will receive a single dose of GSK2239633 or placebo following the standard FDA high fat/high calorie meal. Safety will be monitored (ECGs, telemetry, vital signs, clinical laboratory assessments, adverse events), and blood samples will be taken for pharmacokinetic and pharmacodynamic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with values outside the normal range which are deemed to be clinically relevant should always be excluded from enrollment.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in Section 8.1. This criterion must be followed from the time of the first dose of study medication until 3 months after last dose of study drug.
* Body weight ≥ 50 kg and BMI within the range 18.5-29.9 kg/m2 (inclusive).
* Lifelong non-smokers or ex-smokers of greater than 6 months and < 5 pack year history. Pack years = (cigarettes per day smoked/20) x number of years smoked.
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* Average QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* A positive test for HIV antibody.
* History of alcohol consumption within 6 months of the study defined as:

An average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits.

* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 60 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day or participation in more than 3 clinical studies within 10 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days prior to the first dose of study medication (excluding simple analgesics), unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Urinary cotinine levels indicative of continued smoking or regular use of tobacco- or nicotine-containing products (including snuff, nicotine-containing gum).
* Consumption of grapefruit or grapefruit juice from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-03-29 (Actual); Primary Completion 2011-07-01 (Actual); Study Completion 2011-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GSK2239633 | 0 - 48 hours post dose
  adverse events and clinically relevant changes in safety parameters - 12-lead ECG, telemetry, vital signs (systolic and diastolic blood pressure, heart rate, temperature), clinical laboratory data (haematology, clinical chemistry, urinalysis).

SECONDARY OUTCOMES:
Pharmacokinetics of GSK2239633 | 0 - 48 hours post dose
  Pharmacokinetics: area under the plasma drug concentration versus time curve (AUC(0-t), AUC(0-∞)), maximum observed plasma drug concentration (Cmax), time to maximum observed plasma drug concentration (tmax), apparent clearance (CL/F) and terminal half-life (t1/2) following single oral doses
The relationship between the pharmacokinetics and pharmacodynamics of GSK2239633 | 0 - 48 hours post dose
  Pharmacodynamics: CCR4-mediated T cell actin polymerisation in whole blood
The effect of food on the pharmacokinetics of GSK2239633 | 0 - 24 hours post dose
  Pharmacokinetics: AUC(0-t), Cmax

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Zuidlaren, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Cahn A, Hodgson S, Wilson R, Robertson J, Watson J, Beerahee M, Hughes SC, Young G, Graves R, Hall D, van Marle S, Solari R. Safety, tolerability, pharmacokinetics and pharmacodynamics of GSK2239633, a CC-chemokine receptor 4 antagonist, in healthy male subjects: results from an open-label and from a randomised study. BMC Pharmacol Toxicol. 2013 Feb 28;14:14. doi: 10.1186/2050-6511-14-14. PMID 23448278
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 114660 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/114660?search=study&search_terms=114660#rs
- Available data/document: Annotated Case Report Form: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114660 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register